CLINICAL TRIAL: NCT06082687
Title: De-identified Human Tissue Project for Use with Translational, Biomedical Research At UCF College of Medicine and Burnett School of Biomedical Sciences
Brief Title: De-identified Human Tissue Project
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004397
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Tissue
Keywords: Tissue; surgery; donate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- de-identified human tissue: This Project will receive de-identified human tissue from cooperating institutions for unknown/undisclosed donors.

SUMMARY:
Research scientists of the University of Central Florida College of Medicine (COM) and Burnett School of Biomedical Sciences (BSBS) conduct laboratory studies in biomedical and translational medical research for the purpose of understanding human disease and developing innovative methods for diagnosing, measuring, or treating disease or disease symptoms. The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology.

DETAILED DESCRIPTION:
The objective of this De-Identified Human Tissue Project is the receipt of de-identified human tissue from medical, surgical, and clinical facilities. The human tissue can be fresh or paraffinized. The human tissue will be picked up by the clinical research team and transferred to research scientists of the University of Central Florida's College of Medicine (COM) or Burnett School of Biomedical Sciences (BSBS) for storage and testing according to their separate IRB-approved or IRB-exempted protocols. These separate protocols cannot be for genetic testing. The Project does not receive human tissue resulting from termination of pregnancy.

ELIGIBILITY:
Inclusion:

- de-identified human tissue from cooperating institutions for unknown/undisclosed donors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Not applicable. This Project will receive de-identified human tissue from cooperating institutions for unknown/undisclosed donors.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Receipt of de-identified human tissue for research | 5 years
  The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology. Frequently, these studies require human tissue for testing of assays and devices.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No